CLINICAL TRIAL: NCT02771067
Title: The Utility of Pulse Pressure Variation to Predict the Fluid Responsiveness During Pneumoperitoneum and Reverse-Trendelenburg Position
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 4-2016-0205
Record Dates: First submitted 2016-05-04; First posted 2016-05-12 (Estimated); Last update posted 2017-12-18 (Actual); Status verified 2017-12

CONDITIONS: General Anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pulse pressure variation (Experimental): Pulse pressure variation will be recorded via an arterial catheter after anesthetic induction, before pneumoperitoneum, after pneumoperitoneum, before infusion of 6% hydroxyethyl starch, and after infusion of 6% hydroxyethyl starch. Stroke volume will be also measured to differentiate the fluid responders.
  Interventions: Procedure: Fluid infusion

INTERVENTIONS:
Procedure: Fluid infusion — Fluid infusion will be performed using 6% hydroxyethyl starch. Pulse pressure variation and stroke volume will be measured before and after fluid infusion.

SUMMARY:
The purpose of this study is to investigate the validity of pulse pressure variation to predict fluid responsiveness in patients undergoing robotic or laparoscopic gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

* adult patients aged over 19 years who are scheduled for robotic or laparoscopic gastrectomy

Exclusion Criteria:

* cardiac arrhythmia
* valvular heart disease
* ischemic heart disease
* left ventricular ejection fraction less than 40%
* Pulmonary disease
* esophageal disease
* upper gastrointestinal bleeding
* Body mass index more than 40 kg/m2.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-09-29 (Actual); Primary Completion 2017-02-23 (Actual); Study Completion 2017-02-23 (Actual)

PRIMARY OUTCOMES:
Pulse pressure variation | During the surgery. At Day 0.
  Ability of pulse pressure variation to predict fluid responsiveness will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine Anesthesia and Pain Research Institute Yonsei University, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
The purpose of this study is to investigate the validity of pulse pressure variation to predict fluid responsiveness in patients undergoing robotic or laparoscopic gastrectomy.